CLINICAL TRIAL: NCT02297958
Title: Impact of Fas/FasL in Chemotherapy Response in Epithelial Ovarian Carcinoma
Acronym: IFFaLCCO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01041-46
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Ovarian carcinoma has poor prognosis and new therapeutic strategies are required. Many patients with ovarian carcinoma showed resistance to chemotherapy. Cleaved FasL is known for induced atypical response when is binding to Fas such as avoiding apoptosis and inducing cell motility.

ELIGIBILITY:
Pre-Inclusion Criteria:

- Patient with suspicious ovarian carcinoma using clinical data, biological data (ca125) and radiological data (CT)

Inclusion Criteria:

* Pathological ovarian carcinoma diagnosed at pathological analysis after surgery.
* Neo adjuvant chemotherapy

Exclusion Criteria:

* no neo-adjuvant chemotherapy
* no ovarian carcinoma at final pathological analysis
* less than 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ovarian carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
Correlation between cleaved FasL level ans neoadjuvant chemotherapy tumor response | surgery
  Main outcome is cleaved FasL level and correlation with neoadjuvant chemotherapy tumor response, evaluated during surgery.

SECONDARY OUTCOMES:
Identification of tumoral T cells | surgery
  Identification of tumoral T cells with FACS analysis of dissociated tumor. Different T cells will be studies: Treg/Th17/Th1/Th2 using antibodies against: CD45/CD3/CD4/CD25/FOXP3 (Treg), CD45/CD3/CD4/IL17A (Th17), CD45/CD3/CD4/CD8/IL4/INF (TCD8 and LTCD4 Th1 et Th2).
Disease Free Survival rate | 18 months after surgery
Overall survival rate | 18 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Lavoue, PH, Principal Investigator — Rennes University Hospital
Locations (1):
- Service de Gynécologie, Rennes, France